CLINICAL TRIAL: NCT07247786
Title: Phase II Randomized Clinical Trial for Evaluating the Safety and Feasibility of Fecal Microbiota Transplant (FMT) in Stage II-III Non-small Cell Lung Cancer (NSCLC) Patients, Using Immune Checkpoint Inhibitors (ICI) Responders as Donors.
Brief Title: Study for Evaluating the Safety and Feasibility of Fecal Microbiota Transplant in Stage II-III NSCLC Patients Using ICI Responders as Donors (MIGRANT)
Acronym: MIGRANT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GECP 24/02_MIGRANT; 2025-521251-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Respiratory Tract Neoplasm
Keywords: Non small cell lung cancer; Fecal microbiota transplant; Inmune checkpoint inhibitor responder; Neoadjuvant treatment; Adjuvant treatment; Durvalumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms | interventions — durvalumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Durvalumab + chemotherapy + FMT capsules) (Experimental): The treatment begins with a dose of antibiotics and a fecal microbiota transplant (FMT).
  Neoadjuvant/Induction Treatment:
  Patients will receive intravenous (IV) Durvalumab in combination with IV Paclitaxel and Carboplatin, the latter administered at the end of the Paclitaxel infusion.
  Patients must discontinue study treatment if there is evidence of disease progression that precludes surgery. Patients with stable disease or partial response may still be considered for surgery.
  Surgery:
  After the induction treatment, each patient will be evaluated by a multidisciplinary team at their respective hospital to determine surgical eligibility.
  Adjuvant Treatment:
  Patients with R0 resection confirmed by surgical pathology after surgery will receive adjuvant treatment with IV Durvalumab for several cycles.
  Interventions: Biological: Biological: Fecal Microbiota Transplantation; Drug: Durvalumab; Drug: Paclitaxel; Drug: Carboplatin (AUC 6)
- Control Arm (Durvalumab + chemotherapy) (Active Comparator): Neoadjuvant/Induction Treatment:
  Patients will receive intravenous (IV) Durvalumab in combination with IV Paclitaxel and Carboplatin, the latter administered at the end of the Paclitaxel infusion.
  Patients must discontinue study treatment if there is evidence of disease progression that precludes surgery. Patients with stable disease or partial response may still be considered for surgery.
  Surgery:
  After the induction treatment, each patient will be evaluated by a multidisciplinary team at their respective hospital to determine surgical eligibility.
  Adjuvant Treatment:
  Patients with R0 resection confirmed by surgical pathology after surgery will receive adjuvant treatment with IV Durvalumab for several cycles.
  Interventions: Drug: Durvalumab; Drug: Paclitaxel; Drug: Carboplatin (AUC 6)

INTERVENTIONS:
Biological: Biological: Fecal Microbiota Transplantation — Patients who are going to be donors must have been treated with neoadjuvant chemoimmunotherapy as part of the NADIM studies and must have achieved a pathological complete response (pCR). Additionally, they must be free of disease and complications such as a second tumor or treatment-related toxicity. Samples must be collected from patients who achieved pCR after surgery.
  Patients in the Experimental Arm will receive an antibiotic treatment, followed by the administration of capsules as part of the fecal microbiota transplant (FMT).
  Arms: Experimental Arm (Durvalumab + chemotherapy + FMT capsules)
Drug: Durvalumab — Durvalumab is a human monoclonal antibody of the immunoglobulin G1 kappa (IgG1κ) subclass that inhibits binding of programmed cell death ligand (PD-L1). Durvalumab (MEDI4736) binds with high affinity and specificity to human PD-L1 and blocks its interaction with PD-1 and CD80.
  Pharmaceutical form: Concentrate for solution for infusion (sterile concentrate).Clear to opalescent, colorless to light yellow solution, with no visible particles. The solution has an approximate pH of 6.0 and an osmolality of approximately 400 mOsm/kg.
  Durvalumab will be administered as part of both the neoadjuvant and adjuvant phases of the study.
  Other Names: Imfinzi; MEDI4736
Drug: Paclitaxel — Neoadjuvant / induction treatment: Durvalumab Paclitaxel Carboplatin Neoadjuvant / induction treatment: 4 cycles will be administered prior to the assessment for surgery. Route of administration Paclitaxel: Intravenous infusion. Guidelines of Paclitaxel administration: Paclitaxel must be administered by infusion 200mg/m2 over 3 hours
Drug: Carboplatin (AUC 6) — Neoadjuvant / induction treatment: Durvalumab Paclitaxel Carboplatin* *Infusion at the end of the Paclitaxel infusion. Neoadjuvant / induction treatment 4 cycles will be administered prior to the assessment for surgery. Route of administration Carboplatin: Intravenous infusion. Guidelines of Carboplatin administration: According to the standard of each center.

SUMMARY:
This is a randomized, phase II, multi-centre clinical trial.

Sample size: 68 patients (Experimental Arm (Durvalumab + chemotherapy + FMT capsules): 34 patients, Control Arm (Durvalumab + chemotherapy): 34 patients)

Population: Patients with stage IIA, IIB, IIIA and IIIB (only T3N2) non-small cell lung cancer

In the Experimental arm, patients will receive Fecal Microbiota Transplant. Once done, the patient will start neoadjuvant treatment with Durvalumab + Chemotherapy .

In the Control arm, patients will receive neoadjuvant treatment with Durvalumab + Chemotherapy.

After neoadjuvant/induction treatment every patient will be evaluated to decide if the patient is a candidate for surgery or not. Patients that are R0 after surgery will receive Adjuvant treatment with Durvalumab.

The primary objective is to evaluate the pathological Complete Response (pCR) rate.

The total trial duration will be 6.5 years approximately.

DETAILED DESCRIPTION:
This is a randomized, phase II, multi-centre clinical trial stratified according to PDL1 status (≥50 % or <50%), and Akkermansia positive vs negative.

In the pre-treatment phase, donors will be selected for preparing the fecal microbiota transplant with their samples.

After that, patient's candidate with stage IIA, IIB, IIIA and IIIB (only T3N2) non-small cell lung cancer to study will be randomized in two different arms.

In the Experimental arm, after randomization, patients will receive treatment with Rifaximin. Once done, the patient will start neoadjuvant treatment with Durvalumab IV + Chemotherapy for several cycles.

In the Control arm, after randomization patients will receive neoadjuvant treatment with Durvalumab IV + Chemotherapy for several cycles.

After neoadjuvant/induction treatment every patient will be evaluated by a multidisciplinary team in each participant hospital to decide if the patient is a candidate for surgery or not.

Patients that are R0 confirmed by surgical pathology evaluation after surgery will receive Adjuvant treatment with Durvalumab IV.

Sample size: 68 patients (Experimental Arm (Durvalumab + chemotherapy + FMT capsules): 34 patients, Control Arm (Durvalumab + chemotherapy): 34 patients)

The primary objective is to evaluate the pathological Complete Response (pCR) rate in the intention to treat population (ITT population)

The total trial duration will be 6.5 years approximately.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with histologically- or cytologically- documented NSCLC who present stage IIA, IIB, IIIA or IIIB (only T3N2) disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology)
* PET scan and brain CT or MRI at baseline to confirm the absence of distant disease
* ECOG (Performance status) 0-1
* Adequate hematologic and organ function.
* All patients are notified of the investigational nature of this study and signed a written in-formed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention
* Adequate lung function: Forced Espiratoy Volumen in 1 second (FEV1) >50% of normal volume and Difusion Capacity of the Lungs for Carbon Monoxide (DLCO) >40% of normal value
* Patients aged ≥ 18 years at the time of study entry
* Body weight > 30Kg (for durvalumab monotherapy)
* PDL1 analyzed (value in %)
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective forms of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 6 months after the last dose of trial treatment.
* For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate when used consistently and correctly, and to continue its use for 6 months after the last dose of trial treatment.
* Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drugs. The same rules are valid for male patients involved in this clinical study if they have a partner of childbirth potential. Male patients must always use a condom.
* Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 8 days prior to initiation of study drug.
* Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Presence of at least one measurable lesion by CT-SCAN, as defined by RECIST v1.1.
* Patients with a life expectancy ≥12 weeks.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations

Exclusion Criteria:

* Patients with known sensitizing mutation or an amplification in the epidermal growth factor receptor (EGFR) gene or any variety of alterations of ALK oncogene.
* Known STK-11 ligand alterations, MDM2 amplifications or ROS1 translocations.
* Weight loss >10% within the previous 3 months.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment.
* Patients with other active malignancy requiring concurrent intervention and/or concurrent treatment with other investigational drugs or anti-cancer therapy
* History of active primary immunodeficiency
* History of another primary malignancy.
* Active or prior documented autoimmune or inflammatory disorders.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization.
* Pleural or pericardial effusion.
* Patients who have experienced untreated and/or uncontrolled cardiovascular conditions and/or have symptomatic cardiac dysfunction.
* Positive test for HIV.
* Patients with positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Patients with history of allergy to study drug components/excipients.
* Active tuberculosis.
* Severe infections within 4 weeks prior to be included in the study.
* Major surgical procedure other than for diagnosis within 28 days prior to inclusion or anticipation of need for a major surgical procedure during the course of the study.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.
* Patients with medical, mental, neurological or psychological condition which in the opinion of the investigator would not permit the patient to understand the patient information sheet or comply with study procedures.
* Treatment with any other investigational agent with therapeutic intent within 28 days prior to initiation of study treatment.
* Patients with uncontrolled comorbidities that may affect the clinical trial compliance.
* Women who are pregnant or in the breastfeeding period or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.
* Patients must be informed that they are not allowed to donate blood during the treatment period of this clinical trial.
* Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
* Receipt of a live attenuated vaccine within 30 days prior to the first dose of investigational product (IP).
* Concurrent enrollment in another clinical study, except in cases where the study is observational (non-interventional) or the patient is in the follow-up phase of a previous interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2031-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | From date of randomization until the date of last follow up, assessed up to 24 months
  Pathological Complete Response (pCR) defined as the absence of residual tumor in lung and lymph nodes after surgery.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of last follow up, assessed up to 24 months
  Progression free survival (PFS) defined as the time from initiation of treatment to the occurrence of disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Overall Survival (OS) | From date of randomization until the date of last follow up, assessed up to 24 months
  Overall survival (OS) defined as the time which begins at the start of treatment and up to the time of death or last follow up
Resectability rate (%) | From date of randomization until the date of last follow up, assessed up to 24 months
  Resectability rate defined as the percentage of patients resected divided by the total number of patients who received neoadjuvant treatment
Proportion of R0 resections (%) | From date of randomization until the date of last follow up, assessed up to 24 months
  Percentage of R0 resection will be calculated by dividing the total number of R0 resection patients by the total number of patients resected.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 90 days after the final administration of the drug.]
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — President of Grupo Español de Cáncer de Pulmón
Locations (20):
- Spain (20):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital General Universitario De Elche, Elche, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Quiron Dexeus, Barcelona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada, Granada
  - Complexo Hospitalario Universitario De Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Clinico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario 12 De Octubre, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia, Murcia
  - Hospital Universitario Regional de Málaga, Málaga, Málaga
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital Universitario La Fe, Valencia, Valencia
  - Complexo Hospitalario Universitario De Vigo, Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org